CLINICAL TRIAL: NCT05772156
Title: Prophylactic Methylergonovine in Patients Undergoing Cesarean Delivery With Twin Gestations: A Randomized Controlled Trial
Brief Title: Prophylactic Methylergonovine for Twin Cesarean
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Mirella Mourad, Assistant Professor of Obstetrics and Gynecology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AAAU3902
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Twin; Complicating Pregnancy; Postpartum Hemorrhage
MeSH Terms: conditions — Pregnancy Complications; Postpartum Hemorrhage | interventions — Methylergonovine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prophylactic methylergonovine (Experimental): Prophylactic methylergonovine 200mcg IM
  Interventions: Drug: Methylergonovine
- Control group/placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylergonovine — Methylergonovine 200mcg Intramuscular (IM)
  Other Names: Methergine
  Arms: Prophylactic methylergonovine
Drug: Placebo — Matching saline placebo
  Other Names: Saline
  Arms: Control group/placebo

SUMMARY:
Obstetrical hemorrhage (excessive bleeding related to pregnancy) is a leading cause of maternal morbidity (disease or symptom of disease) and mortality (death) worldwide with a significantly higher frequency and severity following cesarean delivery. Twin gestations (twin pregnancy) are at particularly higher risk for postpartum hemorrhage, yet the management of obstetrical bleeding following twin delivery remains identical to singleton delivery.

The purpose of this study is to understand the effect of prophylactic methylergonovine on blood loss in scheduled twin pregnancy cesarean deliveries. Participants will be randomized (like tossing a coin) to Methylergonovine (investigational drug) or water with salt (saline) (placebo). Methylergonovine or saline will be given as an injection immediately after delivery.

DETAILED DESCRIPTION:
Obstetrical hemorrhage is a leading cause of maternal morbidity and mortality worldwide with a significantly higher frequency and severity following cesarean delivery. In 2020, 31.9 percent of pregnant women in the United States underwent cesarean delivery, making it the second most common operation performed. Though multiple complications can occur following cesarean delivery, hemorrhage morbidities are among the most common with significant cardiovascular implications. Twin gestations are at particularly higher risk for postpartum hemorrhage due to impaired myometrial contractility and atony following overdistention; increased maternal blood volume; and increased uterine blood flow compared to singletons, yet the management of obstetrical bleeding following twin delivery remains identical to singleton delivery. Current strategies to address intrapartum hemorrhage have relied on pharmacological and mechanical treatments after intraoperative identification. However, there is extensive work on prophylactic therapies administered intraoperatively to prevent obstetrical hemorrhage. Recent evidence has emerged about the utility of prophylactic Methylergonovine for the prevention of obstetrical hemorrhage. Methylergonovine, a semisynthetic ergot alkaloid, acts primarily on alpha adrenergic receptors of uterine and vascular smooth muscle, increasing uterine tone and promoting vasoconstriction. In a randomized trial of 80 women undergoing intrapartum cesarean delivery found that fewer patients who were allocated to the methylergonovine group received additional uterotonic agents (20% vs 55%, relative risk (RR) 0.4, 95% confidence interval (CI) 0.2-0.6). Participants receiving methylergonovine were more likely to have satisfactory uterine tone (80% vs 41%, RR 1.9, 95% CI 1.5-2.6), lower incidence of postpartum hemorrhage (35% vs 59%, RR 0.6, 95% CI 0.4-0.9), lower mean quantitative blood loss (967 mL vs 1,315 mL; mean difference 348, 95% CI 124-572), and a lower frequency of blood transfusion (5% vs 23%, RR 0.2, 95% CI 0.1-0.6). Investigators concluded that the administration of prophylactic methylergonovine in addition to oxytocin in patients undergoing intrapartum cesarean birth reduces the need for additional uterotonic agents. In a prospective study of 1210 participants found that intraoperative, prophylactic methylergonovine decreased post-operative blood loss with no adverse side effects. Randomized trials of Methylergonovine as prophylaxis to prevent hemorrhage in cesarean delivery have exclude twin gestations. Currently, there remains a paucity of research regarding prophylactic procedures for twin cesarean delivery. There is an opportunity to prophylactically address hemorrhage in high-risk groups. Therefore, the investigators propose a prospective randomized controlled trial which will compare maternal blood loss associated with prophylactic methylergonovine during cesarean delivery among patients with twin.

ELIGIBILITY:
Inclusion Criteria:

* Twin gestation
* Scheduled cesarean delivery (>=34 weeks)

Exclusion criteria:

* Patients with known hypertensive disease: history of chronic hypertension, gestational hypertension or preeclampsia with or without severe features
* Use of protease inhibitors given known vasoconstrictive side effects with concomitant methylergonovine administration
* Hypersensitivity to methylergonovine or any of the ingredients
* Participating in another intervention study where the primary outcome includes postpartum bleeding or thromboembolism, or the study intervention directly affects postpartum bleeding or thromboembolism
* Receipt of uterotonics, other than oxytocin, or planned or expected use of uterotonic prophylaxis
* Non-elective cesarean delivery

Max Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mirella Mourad, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is currently undecided if the Individual participant data (IPD) will be shared.
  If there is a plan to share the following will be shared: the IPD that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices), the Study Protocol, Statistical Analysis Plan, and, Informed Consent Form documents. The timeframe for which the IPD will be shared is beginning 3 months and ending 5 years following article publication. Data will be shared with researchers who provide a methodologically sound proposal, so that they may achieve aims in the proposal.

REFERENCES:
- [Background] Osterman M, Hamilton B, Martin JA, Driscoll AK, Valenzuela CP. Births: Final Data for 2020. Natl Vital Stat Rep. 2021 Feb;70(17):1-50. PMID 35157571
- [Background] Sheehan SR, Montgomery AA, Carey M, McAuliffe FM, Eogan M, Gleeson R, Geary M, Murphy DJ; ECSSIT Study Group. Oxytocin bolus versus oxytocin bolus and infusion for control of blood loss at elective caesarean section: double blind, placebo controlled, randomised trial. BMJ. 2011 Aug 1;343:d4661. doi: 10.1136/bmj.d4661. PMID 21807773
- [Background] Blitz MJ, Yukhayev A, Pachtman SL, Reisner J, Moses D, Sison CP, Greenberg M, Rochelson B. Twin pregnancy and risk of postpartum hemorrhage. J Matern Fetal Neonatal Med. 2020 Nov;33(22):3740-3745. doi: 10.1080/14767058.2019.1583736. Epub 2019 Mar 5. PMID 30836810
- [Background] Attilakos G, Psaroudakis D, Ash J, Buchanan R, Winter C, Donald F, Hunt LP, Draycott T. Carbetocin versus oxytocin for the prevention of postpartum haemorrhage following caesarean section: the results of a double-blind randomised trial. BJOG. 2010 Jul;117(8):929-36. doi: 10.1111/j.1471-0528.2010.02585.x. Epub 2010 May 19. PMID 20482535
- [Background] Chaudhuri P, Banerjee GB, Mandal A. Rectally administered misoprostol versus intravenous oxytocin infusion during cesarean delivery to reduce intraoperative and postoperative blood loss. Int J Gynaecol Obstet. 2010 Apr;109(1):25-9. doi: 10.1016/j.ijgo.2009.11.009. Epub 2010 Jan 13. PMID 20070961
- [Background] Senturk S, Kagitci M, Balik G, Arslan H, Kir Sahin F. The Effect of the Combined Use of Methylergonovine and Oxytocin during Caesarean Section in the Prevention of Post-partum Haemorrhage. Basic Clin Pharmacol Toxicol. 2016 May;118(5):338-43. doi: 10.1111/bcpt.12500. Epub 2015 Nov 15. PMID 26449959
- [Background] Masse N, Dexter F, Wong CA. Prophylactic Methylergonovine and Oxytocin Compared With Oxytocin Alone in Patients Undergoing Intrapartum Cesarean Birth: A Randomized Controlled Trial. Obstet Gynecol. 2022 Aug 1;140(2):181-186. doi: 10.1097/AOG.0000000000004857. Epub 2022 Jul 6. PMID 35852267
- [Background] Horowitz E, Yogev Y, Ben-Haroush A, Rabinerson D, Feldberg D, Kaplan B. Routine hemoglobin testing following an elective Cesarean section: is it necessary? J Matern Fetal Neonatal Med. 2003 Oct;14(4):223-5. doi: 10.1080/jmf.14.4.223.225. PMID 14738165

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Normal Saline 1mL
Period: Overall Study
Arm/Group | Prophylactic Methylergonovine | Placebo
Started | 33 | 33
Completed | 33 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylactic Methylergonovine | Placebo | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 33 | 66
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 9 | 20
  White | 22 | 22 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 14 | 29
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown or Not Reported | 0 | 0 | 0
Number of Prior Cesarean Deliveries, n (%) [Count of Participants; unit: Participants]
  0 | 23 | 24 | 47
  1 | 7 | 7 | 14
  >=2 | 3 | 2 | 5
Chorionicity, n (%) [Count of Participants; unit: Participants]
  Dichorionic | 21 | 21 | 42
  Monochorionic-Diamniotic | 12 | 12 | 24
Maternal BMI (kg/m2), mean, SD [Mean (Standard Deviation); unit: kg/m^2] | 30.0 (5.7) | 30.5 (7.3) | 30.25 (6.5)
Tobacco use in pregnancy, n (%) [Count of Participants; unit: Participants] | 1 | 0 | 1
Gestational diabetes mellitus, n (%) [Count of Participants; unit: Participants] | 5 | 6 | 11
Preoperative maternal hemoglobin level (g/dL), mean (SD) [Mean (Standard Deviation); unit: g/dL] | 11.6 (1.2) | 12.0 (1.3) | 11.8 (1.25)

OUTCOME MEASURES:

1. Primary Outcome: Change in Maternal Hemoglobin Level
Description: The change in maternal hemoglobin level as taken from blood samples. The change will be calculated from preoperative day 1 (baseline) to postoperative day 1.
Time Frame: Baseline and Postoperative Day 1 (Approximately 48 hours)
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Placebo Group: Normal Saline 1mL
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
g/dL | 1.1 (0.7) | 2.1 (0.9)

2. Secondary Outcome: Surgical Time
Description: Surgical time measured from the time of incision to closure
Time Frame: Intraoperative (Approximately 24 hours)
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
Minutes | 62.0 [54 to 75] | 61.0 [49 to 69]

3. Secondary Outcome: Estimated Blood Loss
Description: At the end of the surgery, the primary surgeon will estimate the blood loss throughout the case.
Time Frame: Intraoperative (Approximately 24 hours)
Measure: Median (Inter-Quartile Range); unit: cc
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
cc | 800 [800 to 900] | 1000 [800 to 1098]

4. Secondary Outcome: Quantitative Blood Loss
Description: Quantitative blood loss is calculated by weighing the used towels during the operation. The number is calculated by the circulating nurse in the operating room.
Time Frame: Intraoperative (Approximately 24 hours)
Measure: Median (Inter-Quartile Range); unit: cc
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
cc | 891 [743 to 966] | 1017 [931 to 1211]

5. Secondary Outcome: Number of Participants With Postpartum Hemorrhage
Description: The number of participants with postpartum hemorrhage (defined as estimated blood loss >1000 cc)
Time Frame: Intraoperative (Approximately 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
Participants | 6 | 18

6. Secondary Outcome: Number of Participants Requiring Use of Uterotonics
Description: Number of participants given uterotonics, such as prostaglandins
Time Frame: Intraoperative (Approximately 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
Participants | 0 | 6

7. Secondary Outcome: Number of Participants Requiring Use of Tranexamic Acid
Description: Number of participants given Tranexamic acid
Time Frame: Intraoperative (Approximately 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
Participants | 2 | 7

8. Secondary Outcome: Number of Participants Requiring Use of Open-Label Methylergonovine
Description: Number of participants requiring the use of any amount of open-label methylergonovine (not blinded study drug)
Time Frame: Intraoperative (Approximately 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
Participants | 0 | 7

9. Secondary Outcome: Number of Participants Requiring Transfusion (Intraoperative)
Description: Number of participants requiring transfusion of 1 or more units of packed red blood cells, including whole blood or cell saver.
Time Frame: Intraoperative (Approximately 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Surgical or Radiological Interventions
Description: Composite number of surgical or radiological interventions (such as: laparotomy, evacuation of hematoma, hysterectomy, uterine packing, intrauterine balloon tamponade, interventional radiology) to control bleeding and related complications or maternal death.
Time Frame: Intraoperative (Approximately 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Transfusion Related Acute Lung Injury (TRALI)
Description: Number of participants with transfusion related acute lung injury (TRALI)
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
Participants | 0 | 0

12. Secondary Outcome: Number of Participants Requiring Transfusion (6 Weeks)
Description: Number of participants requiring transfusion of 1 or more units of fresh frozen plasma, cryoprecipitate, or platelets or administration of any factor concentrates.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
Participants | 2 | 4

13. Secondary Outcome: Number of Participants With Acute Elevation of Serum Creatinine
Description: Number of participants with acute elevation of serum creatinine of ≥ 0.3 mg/dL
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
Participants | 0 | 0

14. Secondary Outcome: Number of Postpartum Infectious Complications
Description: Number of Postpartum infectious complications such as: endometritis, surgical site infection, pelvic abscess
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
Participants | 0 | 2

15. Secondary Outcome: Number of Participants With Admission to the Intensive Care Unit
Description: Number of participants with admission to the intensive care unit for more than 24 hours
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
Participants | 0 | 0

16. Secondary Outcome: Length of Stay
Description: Length of stay measured from the time of hospital admission to hospital discharge.
Time Frame: Up to 6 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
days | 4 [3 to 4] | 4 [4 to 6]

17. Secondary Outcome: Number of Participants Re-Admitted to the Hospital
Description: The number of participants who experienced hospital re-admission
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 33 | 33
Participants | 1 | 3

18. Secondary Outcome: Apgar Scores
Description: Apgar score is a measure of the physical condition of a newborn infant. Scores range from 0-10 with a higher score indicating a better outcome; Apgar score of 0-3 is low, 4-6 is moderately abnormal, and 7-10 is reassuring.
Time Frame: 1 and 5 minutes post-delivery (approximately 24 hours post-baseline)
Population: Newborns were assessed rather than the mothers (i.e. enrolled participants). Each participant gave birth to twins (66 newborns total). Newborns were not considered enrolled but did contribute to this assessment.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 66 | 66
score on a scale
  Apgar 1 minute | 8 [8 to 9] | 8 [8 to 8]
  Apgar 5 minutes | 9 [9 to 9] | 9 [9 to 9]

19. Secondary Outcome: Neonatal Intensive Care Unit (NICU) Admission
Description: Number of newborns admitted to the neonatal intensive care unit (NICU).
Time Frame: Time of delivery (Approximately 24 hours)
Population: as for outcome 18
Measure: Number; unit: newborns
Arm/Group | Prophylactic Methylergonovine | Placebo Group
Number analyzed (Participants) | 66 | 66
newborns | 19 | 20

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 6 weeks
Arm/Group | Prophylactic Methylergonovine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT05772156/Prot_SAP_000.pdf